CLINICAL TRIAL: NCT00189696
Title: Phase 3 Study of YM060 in Patients With Diarrhea-predominant Irritable Bowel Syndrome (d-IBS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 060-CL-202
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome, Diarrhea
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea | interventions — ramosetron

INTERVENTIONS:
Drug: YM060

SUMMARY:
This study will examine the efficacy, safety and tolerability of oral dose of YM060, 5-HT3 receptor antagonist, in patients with d-IBS.

ELIGIBILITY:
Inclusion Criteria:

* Patients satisfying the Rome II Diagnostic Criteria.
* Patients in whom no organic changes were observed in large intestine.

Exclusion Criteria:

* Patients have diseases which interfere with evaluation of the efficacy and safety in this study.
* Patients are receiving and/or have received prior to the enrollment the treatment which interfere with evaluation of the efficacy and safety in this study.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Clinical Development III, Study Chair — Astellas Pharma Inc
Locations (4):
- Japan (4):
  - Chubu Region
  - Kanto Region
  - Shikoku Region
  - Tohoku Region

REFERENCES:
- [Background] Matsueda K, Harasawa S, Hongo M, Hiwatashi N, Sasaki D. A randomized, double-blind, placebo-controlled clinical trial of the effectiveness of the novel serotonin type 3 receptor antagonist ramosetron in both male and female Japanese patients with diarrhea-predominant irritable bowel syndrome. Scand J Gastroenterol. 2008;43(10):1202-11. doi: 10.1080/00365520802240255. PMID 18618371
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=060-CL-202